CLINICAL TRIAL: NCT00636259
Title: A Compassionate Use Trial With Bicalutamide (Casodex) 150-mg for Subjects With Prostate Cancer
Brief Title: Casodex 150-mg Compassionate Use Trial for Subjects With Prostate Cancer
Status: No longer available | Type: Expanded Access
Sponsor: AstraZeneca (Industry)
Other Study IDs: 7054US/0014; D6874L00006
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2008-06-11 (Estimated); Status verified 2008-06

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: Prostate cancer; Casodex
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide

INTERVENTIONS:
Drug: Bicalutamide (Casodex) — 150mg

SUMMARY:
This study provides compassionate use of bicalutamide (Casodex) at a 150-mg dose for subjects with prostate cancer prior to it becoming commercially available. The patient will receive bicalutamide 150-mg as long as the physician feels that the subject is benefiting from this therapy and safety information is provided regularly to AstraZeneca. Treatment will be discontinued after bicalutamide 150-mg becomes commercially available.

ELIGIBILITY:
Inclusion Criteria:

* Patients with adenocarcinoma of the prostate
* Subjects with locally advanced, and/or metastatic prostate cancer for whom surgical castration or other medical interventions are not considered appropriate or acceptable

Exclusion Criteria:

* Any known history of abnormal liver function tests
* Any severe concomitant condition that would make it undesirable, in the clinician's opinion, for the subject to participate in the trial.
* Known hypersensitivity to bicalutamide or any of the components found in bicalutamide

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult